CLINICAL TRIAL: NCT04958239
Title: An Open Label, Phase I Dose-finding and Expansion Study of BI 765179 as Monotherapy and in Combination With Ezabenlimab (BI 754091) in Patients With Advanced Solid Cancers, and BI 765179 in Combination With Pembrolizumab in First-line PD-L1-positive Metastatic or Incurable, Recurrent Head and Neck Squamous Cell Carcinoma (HNSCC)
Brief Title: A Study to Test BI 765179 Alone and in Combination With Ezabenlimab in Patients With Advanced Cancer (Solid Tumors) and BI 765179 in Combination With Pembrolizumab in Patients With Advanced Head and Neck Cancer
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1463-0001; 2021-000234-34 (EudraCT Number); 2023-510307-22-00 (Registry Identifier: CTIS (EU)); U1111-1310-6376 (Registry Identifier: WHO International Clinical Trials Registry Platform (ICTRP))
Record Dates: First submitted 2021-07-01; First posted 2021-07-12 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2026-02

CONDITIONS: Neoplasms
MeSH Terms: conditions — Neoplasms | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 1 Arm A: BI 765179 (Experimental)
  Interventions: Drug: BI 765179
- Phase 1a Arm B: BI 765179 + ezabenlimab (Experimental)
  Interventions: Drug: BI 765179; Drug: Ezabenlimab
- Phase 1b Cohort 1: pembrolizumab + low dose of BI 765179 (Experimental)
  Interventions: Drug: BI 765179; Drug: Pembrolizumab
- Phase 1b Cohort 2: pembrolizumab + high dose of BI 765179 (Experimental)
  Interventions: Drug: BI 765179; Drug: Pembrolizumab

INTERVENTIONS:
Drug: BI 765179 — BI 765179
Drug: Ezabenlimab — Ezabenlimab
  Arms: Phase 1a Arm B: BI 765179 + ezabenlimab
Drug: Pembrolizumab — Pembrolizumab
  Arms: Phase 1b Cohort 1: pembrolizumab + low dose of BI 765179; Phase 1b Cohort 2: pembrolizumab + high dose of BI 765179

SUMMARY:
This study is open to adults with advanced cancer (solid tumors) and people with advanced head and neck cancer. The study has 2 parts. The purpose of Part 1 of this study is to find the highest dose of a medicine called BI 765179 that people with solid tumors can tolerate when taken alone or together with a medicine called ezabenlimab. The goal of Part 2 is to find out whether BI 765179 in combination with a medicine called pembrolizumab helps people with advanced head and neck cancer.

In Part 1, each participant is put into 1 of 2 groups. Participants get BI 765179 alone or in combination with ezabenlimab as infusion into a vein every 3 weeks. In Part 2, participants are also divided into 2 groups. 1 group gets a low dose of BI 765179 in combination with pembrolizumab and the other group gets a high dose of BI 765179 in combination with pembrolizumab. Participants receive the study treatment as infusions into a vein.

BI 765179, ezabenlimab, and pembrolizumab are antibodies that may help the immune system fight cancer. In this study, BI 765179 is given to people for the first time.

Participants can stay in the study up to 2 years if they benefit from treatment and can tolerate it. The doctors regularly check the participants' health and note any health problems that could have been caused by the study treatment.

ELIGIBILITY:
Inclusion Criteria:

All cohorts:

* Patients with locally advanced, unresectable or metastatic solid tumors who are either refractory after standard therapy for the disease or for whom standard therapy is not appropriate
* Tumor with expected high expression of Fibroblast activation protein (FAP) of the following histologies:

  * Non-small cell lung carcinoma (NSCLC)
  * Gastric cancer
  * Esophageal adenocarcinoma or squamous cell carcinoma
  * Urothelial bladder carcinoma
  * Head and neck squamous cell carcinoma
  * Cutaneous malignant melanoma
  * Cutaneous squamous cell carcinoma
  * Hepatocellular carcinoma
  * Pancreatic adenocarcinoma
  * Colorectal cancer
  * Malignant pleural mesothelioma
  * Cervical squamous cell cancer
  * Ovarian carcinoma
  * Triple-negative breast cancer
* At least 18 years of age at the time of the consent or over the legal age of consent in countries where that is greater than 18 years
* Signed and dated, written informed consent (IC) in accordance with ICH-GCP and local legislation prior to admission to the trial
* At least one measurable lesion outside of central nervous system (CNS) as defined per modified Response evaluation criteria in solid tumors (RECIST) v1.1
* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Adequate liver, bone marrow and renal organ function
* Male or female patients. Women of childbearing potential (WOCBP) and men able to father a child must be ready and able to use highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. These methods must be used during the study and for at least 6 months after the last dose of the study medication. A list of contraception methods meeting these criteria is provided in the patient information.
* Patients with brain metastases are eligible provided they meet all of the following criteria:

  * Brain metastases have adequately been treated and are considered stable by the Investigator
  * Radiotherapy or surgery for brain metastases was completed at least 2 weeks prior to the first administration of BI 765179
  * Patient is off steroids for at least 7 days (physiologic doses of steroids is permitted, if this was stable for the last 4 weeks)
  * The patient is off anti-epileptic drugs for at least 7 days

Back-fill cohorts only:

* Patient has agreed to and signed an IC form to provide mandatory pre-treatment and on-treatment fresh tumor biopsy
* At least one lesion (separate from the evaluable target lesion outside of the CNS as defined per RECIST v1.1) that is accessible for mandatory paired pre and on-treatment biopsy

Phase 1b:

* Histologically or cytologically confirmed diagnosis of metastatic or incurable, recurrent head and neck squamous cell carcinoma (HNSCC)
* No prior systemic therapy administered in the metastatic or incurable, recurrent setting
* Primary tumor locations of oropharynx, oral cavity, hypopharynx, or larynx
* At least 18 years of age at the time of the consent or over the legal age of consent in countries where that is greater than 18 years
* Signed and dated written IC in accordance with ICH-GCP and local legislation prior to admission to the trial Further inclusion criteria apply

Exclusion Criteria:

Phase 1a

* Currently enrolled in another investigational device or drug trial
* Previous or concomitant malignancies other than the one treated in this trial within the last 2 years except:

  * Effectively treated non-melanoma skin cancers
  * Effectively treated carcinoma in situ of the cervix
  * Effectively treated ductal carcinoma in situ
  * Other effectively treated malignancy that is considered cured by 'local treatment'
* Previous treatment with agents targeting CD137
* Known leptomeningeal disease or spinal cord compression due to disease
* Anticoagulant treatment that cannot be safely interrupted if medically needed (e.g., biopsy) based on the opinion of the Investigator
* Persistent toxicity from previous treatments that has not resolved to ≤ Common terminology criteria for adverse events (CTCAE) Grade 1 (except for alopecia, CTCAE Grade 2 neuropathy, asthenia/fatigue or grade 2 endocrinopathies controlled by replacement therapy)
* Patient has a diagnosis of immunodeficiency
* Patient with history of immunosuppressive medication within 14 days prior to the first dose of BI 765179. The following are exceptions to this criterion:

  * Use of intranasal, inhaled, or topical corticosteroids, local steroid injections (e.g., intra-articular injections)
  * Systemic corticosteroids at physiologic doses ≤10 mg/day (prednisone or equivalent)
  * Physiological replacement dose of corticosteroids Further exclusion criteria apply.

Phase Ib

* Disease suitable for local therapy administered with curative intent
* Participants must not have a primary tumor site of nasopharynx or sino-nasal cancer or salivary gland cancers (any histology)
* Currently enrolled in another investigational device or drug trial
* Life expectancy of <3 months and/or has rapidly progressing disease
* Diagnosed and/or treated additional malignancy within 2 years prior to randomization with the exception of curatively treated basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or curatively resected in situ cervical and/or in situ breast cancers Further exclusion criteria apply

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 149 (Actual)
Dates: Start 2021-10-18 (Actual); Primary Completion 2026-04-29 (Estimated); Study Completion 2028-02-17 (Estimated)

PRIMARY OUTCOMES:
Phase 1a: Maximum Tolerated Dose (MTD) | Up to Day 21 (end of Cycle 1)
  MTD is defined as the highest dose with less than 25% risk of the true Dose Limiting Toxicity (DLT) rate being equal to or above 33% during the MTD evaluation period. The MTD will be assessed based on the number of patients experiencing DLTs, graded according to Common terminology criteria for adverse events (CTCAE) version 5.0, during the MTD evaluation period.
Phase 1a: Occurrence of Dose Limiting Toxicities (DLTs) in the MTD evaluation period | Up to Day 21 (end of Cycle 1)
Phase 1b: Objective response (OR) | Up to 2 years.
  OR is defined as a best overall response of confirmed complete response (CR) or confirmed partial response (PR) according to Response evaluation criteria in solid tumors (RECIST) version (v) 1.1 by Investigator assessment from the date of treatment start until the earliest date of disease progression, death, or last evaluable tumor assessment before start of subsequent anti-cancer therapy, loss to follow-up, or withdrawal of consent.

SECONDARY OUTCOMES:
Phase 1a: Occurrence of DLTs during the on-treatment period (per arm) | up to 36 months
Phase 1a: Maximum measured concentration of BI 765179 in plasma (Cmax) | Up to Day 21 (end of Cycle 1)
Phase 1a: Area under the concentration-time curve of BI 765179 in plasma over a uniform dosing interval from zero to 504h (AUC0-504) | Up to Day 21 (end of Cycle 1)
Phase Ib: Occurrence of adverse events (AEs) using the US National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5 | Up to 2 years.
Phase 1b: Occurrence of serious AEs (SAEs) during the on-treatment period | Up to 2 years.
Phase 1b: OR assessed by the Investigator according to immune-related RECIST (iRECIST) | Up to 2 years.
  OR assessed by the Investigator according to immuno-related RECIST (iRECIST) is defined as best overall response of immune-related complete response (iCR) and immune related partial response (iPR), where the best overall response is the best time point response recorded from the first administration of study medication until the end of treatment.
Phase Ib: Duration of response (DoR) assessed by RECIST v1.1 | Up to 2 years.
  DoR assessed by RECIST v1.1 is defined as the time from first documented CR or PR until the earliest of PD or death among patients with an OR.
Phase 1b: DoR assessed by iRECIST | Up to 2 years.
  DoR assessed by iRECIST is defined as the time from first documented iCR or iPR until the earliest of unconfirmed progression of disease (iUPD) or death among patients with an OR (iCR, iPR).
Phase 1b: Progression-free survival (PFS) in all patients assessed by the Investigator according to RECIST v1.1 | Up to 2 years.
  PFS in all patients assessed by the Investigator according to RECIST v1.1 is defined as the time from first treatment administration until tumor progression or death from any cause, whichever occurs earlier.
Phase 1b: PFS in all patients assessed by the Investigator according to iRECIST | Up to 2 years.
  PFS in all patients assessed by the Investigator according to iRECIST is defined as the time from first administration of study medication until the first date of iUPD (provided that confirmed progressive disease (iCPD) is the next time point response, i.e., progression is confirmed at the next tumor assessment) or death from any cause, whichever occurs earlier.
Phase 1b: PFS rate at 14 weeks | Up to 2 years.
  PFS rate at 14 weeks is defined as the proportion of patients who survive and are progression free at least 14 weeks after the date of first treatment.
Phase 1b: Overall survival (OS) | Up to 2 years.
  OS is defined as the time from first treatment administration until death from any cause.
Phase 1b: OS rate at 12 months | Up to 2 years.
  OS rate at 12 months is defined as the proportion of patients with OS ≥12 months after the date of first treatment.

CONTACTS AND LOCATIONS:
Locations (48):
- United States (5):
  - University of Arizona, Tucson, Arizona
  - Beverly Hills Cancer Center, Beverly Hills, California
  - The University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Avera Cancer Institute, Sioux Falls, South Dakota
  - NEXT Oncology-San Antonio-65273, San Antonio, Texas
- Australia (4):
  - Border Cancer Hospital, Albury, New South Wales
  - Kinghorn Cancer Centre, Darlinghurst, New South Wales
  - Townsville Hospital, Douglas, Queensland
  - Austin Hospital, Heidelberg, Victoria
- Belgium (3):
  - Cliniques Universitaires Saint-Luc, Brussels
  - Edegem - UNIV UZ Antwerpen, Edegem
  - AZ Groeninge, Kortrijk
- Brazil (3):
  - ICESP - Instituto do Cancer do Estado de Sao Paulo, São Paulo
  - Hospital Sírio Libanês-São Paulo-68088, São Paulo
  - Beneficência Portuguesa - Real e Benemérita Associação Portuguesa de Beneficência, São Paulo
- China (5):
  - The First Affiliated Hospital Of Bengbu Medical College, Bengbu
  - Hunan Province Tumor Hospital, Changsha
  - Fujian Cancer Hospital, Fuzhou
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou
  - Wuhan Union Hospital, Wuhan
- Masaryk Memorial Cancer Institute, Brno, Czechia
- France (3):
  - HOP Saint-André, Bordeaux
  - CTR Georges-François Leclerc, Dijon
  - INS Cancérologie Ouest Saint-Herblain, Saint-Herblain
- Germany (3):
  - Universitätsklinikum Freiburg, Freiburg im Breisgau
  - Martin-Luther-Universität Halle-Wittenberg, Halle
  - Klinikum Stuttgart, Stuttgart
- Israel (2):
  - Shaare-Zedek Medical Center, Oncology Institute, Jerusalem
  - Sourasky Medical Center, Tel Aviv
- Istituto Nazionale IRCCS Tumori Fondazione Pascale, Napoli, Italy
- Japan (5):
  - Aichi Cancer Center Hospital, Aichi, Nagoya
  - National Cancer Center Hospital East, Chiba, Kashiwa
  - Kanagawa Cancer Center, Kanagawa, Yokohama
  - Kansai Medical University Hospital, Osaka, Hirakata
  - Osaka International Cancer Institute, Osaka, Osaka
- Mexico (4):
  - Centro Oncologico Internacional, Mexico City
  - Instituto Nacional de Cancerologia, México
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
  - Fundación Santos y de la Garza Evia, I.B.P, Monterrey
- Netherlands (2):
  - VU University Medical Center, Amsterdam
  - Erasmus Medisch Centrum-ROTTERDAM-50697, Rotterdam
- South Korea (3):
  - Gachon University Gil Medical Center, Incheon
  - CHA Bundang Medical Center, Seongnam
  - Asan Medical Center, Seoul
- Spain (4):
  - Hospital Germans Trias i Pujol, Badalona
  - Hospital Universitari Vall D Hebron, Barcelona
  - Hospital Clínico San Carlos, Madrid
  - Clínica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No
Clinical studies sponsored by Boehringer Ingelheim, phases I to IV, interventional and non-interventional, are in scope for sharing of the raw clinical study data and clinical study documents, except for the following exclusions:
  1. studies in products where Boehringer Ingelheim is not the license holder;
  2. studies regarding pharmaceutical formulations and associated analytical methods, and studies pertinent to pharmacokinetics using human biomaterials;
  3. studies conducted in a single center or targeting rare diseases (because of limitations with anonymization).
  For more details refer to: https://www.clinicalstudies.boehringer-ingelheim.com/msw/datasharing

REFERENCES:
- See also: Related Info — http://www.mystudywindow.com